CLINICAL TRIAL: NCT03684863
Title: Randomised, Multicenter Phase II Study in Patients With HER-2 Positive Breast Cancer With Capecitabine Versus Observation With Pathologic Residual Tumors After Preoperative Chemotherapy
Brief Title: Capecitabine in HER-2 Positive Breast Cancer With Pathologic Residual Tumors After Preoperative Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Director of the Breast Surgery Ⅰ, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-06
Record Dates: First submitted 2018-08-26; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy (No Intervention)
- capecitabine (Experimental)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — observation
  Arms: capecitabine

SUMMARY:
This study is designed to investigate the efficacy and safety of capecitabine, as a postoperative adjuvant chemotherapy, for HER-2 positive breast cancer patients who have pathologic residual cancer cells after the preoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with primary, infiltrative breast cancer who has been diagnosed on a histological basis.
2. Stage I-IIIB at the first diagnosis and underwent curative resection.
3. The patient was non-pCR after preoperative chemotherapy including anthracycline agents; that is, she had undergone primary tumor resection and pathologically confirmed to have residual cancer cells. The previously adminstered preoperative chemotherapy must have involved at least four cycles of anthracycline agents. However, even if anthracycline regimen is shorter than 4 courses, the following regimen can be registered.

   * FEC 3 courses (EPI>=100mg/m2)+Docetaxel 3 courses and trastuzumab 3 courses.
   * TCH only over 6 courses
4. The patient has been confirmed to be HER2 positive. etc.
5. The patient's general performance status is 0 to 1.
6. The patient must have no carry-over of efficacy from any previous treatment.
7. The patient has maintained sufficient organ function to permit valid evaluation.
8. The patient must have no adverse drug reactions of grade 2 or higher carried over from previous treatment.
9. The patient's creatinine clearance is higher than 50 ml/min
10. The patient has personally given written, informed consent to participate in this study.

Exclusion Criteria:

1. The patient is considered to require postoperative chemotherapy other than capecitabine.
2. The patient has previously been treated with oral 5-FU agents (however, previous treatment with iv 5-FU is acceptable).
3. The patient has either simultaneous or non-simultaneous bilateral breast cancer.
4. The patient has a history of other malignancies or synchronic multiple cancers. However, lesions corresponding to carcinoma in situ or intramucosal carcinoma healed by topical therapy are eligible.
5. The patient is pregnant, has the potential and/or wishes to become pregnant, or is breastfeeding.
6. The patient has previously had an organ transplant.
7. The patient shows hypersensitivity to fluoropyrimidine agents; has previously suffered severe adverse drug reactions with fluoropyrimidine agents; or has a history of serious hypersensitivity to LHRH analogs, tamoxifen, letrozole, anastrozole, and/or exemestane.
8. The patient is currently suffering from serious complications or associated disorders, such as malignant hypertension, congestive heart failure, coronary failure, arrhythmias requiring treatment, infectious diseases, and/or hemorrhagic tendency, and/or has suffered a myocardial infarction within the previous 6 months.
9. The patient has a fever, and there is the possibility that she has an infection.
10. The patient has been shown to have metastasis to other organs.
11. The patient requires treatment for epilepsy and/or central nervous system disorders.
12. The patient is currently being treated for, or has a history of, psychiatric disease.
13. It would be difficult to orally administer drugs to the patient, and/or she suffers from functional insufficiency of the upper gastrointestinal tract and/or malabsorption syndrome.
14. For any other reason, the investigator or sub-investigator has judged the patient to be ineligible for participation.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival(DFS) | 5 years
  To determine the percentage of disease-free survival (DFS) for the capecitabine monotherapy arm or placebo arm.

SECONDARY OUTCOMES:
overall survival(OS) | 5 years
  To determine the percentage of disease-free survival (DFS) for the capecitabine monotherapy arm or placebo arm.
medicine safety | 5 years
  To determine the percentage of disease-free survival (DFS) for the capecitabine monotherapy arm or placebo arm.